CLINICAL TRIAL: NCT05133167
Title: Comparison of Efficacy of Surgical Interventions (Balloon Tamponade Versus B-lynch Suture) to Prevent Postpartum Hemorrhage in Patients With Placenta Previa
Brief Title: Balloon Tamponade Vs B-Lynch In Placenta Previa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CMH Jhelum (Other)
Responsible Party: Principal Investigator, M. Awais Qarni, Anesthesiologist, CMH Jhelum
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16112021
Record Dates: First submitted 2021-11-15; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-04

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa | interventions — Balloon Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Experimental): In group A, balloon tamponade (using Foley catheter 28 Fr) was used intra-operatively to prevent post-partum hemorrhage.
  Interventions: Procedure: Balloon Tamponade or B-Lynch
- GROUP B (Experimental): In group B, B lynch suture was used intra-operatively to prevent post-partum hemorrhage.
  Interventions: Procedure: Balloon Tamponade or B-Lynch

INTERVENTIONS:
Procedure: Balloon Tamponade or B-Lynch — In group A, balloon tamponade (using Foley catheter 28 Fr) was used intra-operatively to prevent post-partum hemorrhage. Post-operative blood loss within first 24 hours was estimated by measuring the amount of blood collected in Foley balloon tamponade bag, in milliliters. In group B, B lynch suture was used intra-operatively to prevent post-partum hemorrhage. Post-operative blood loss within first 24 hours was estimated by the weight difference of the pads before and after patient use (1-gram weight difference = 1 ml blood volume lost). Mean blood loss within first 24 hours post procedure, was compared in both the groups for outcome measurement.

SUMMARY:
Patients were allocated to group A and B. In group A, balloon tamponade (using Foley catheter 28 Fr) was used intra-operatively to prevent post-partum hemorrhage. In group B, B lynch suture was used intra-operatively to prevent post-partum hemorrhage.

DETAILED DESCRIPTION:
After approval from hospital ethical committee, patients fulfilling the inclusion & exclusion criteria were recruited after taking informed written consent for surgery. Patients were allocated to group A and B using computer generated random sample allocation.

In group A, balloon tamponade (using Foley catheter 28 Fr) was used intra-operatively to prevent post-partum hemorrhage. Post-operative blood loss within first 24 hours was estimated by measuring the amount of blood collected in Foley balloon tamponade bag, in milliliters.

In group B, B-lynch suture was used intra-operatively to prevent post-partum hemorrhage. Post-operative blood loss within first 24 hours was estimated by the weight difference of the pads before and after patient use (1-gram weight difference = 1 ml blood volume lost). Mean blood loss within first 24 hours post procedure, was compared in both the groups for outcome measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton pregnancy
2. Late Third Trimester pregnancy (35+ weeks to 39 weeks)
3. Placenta Previa confirmed by ultrasonography
4. Elective Caesarean Section.

Exclusion Criteria:

1. Multiple gestation
2. Placenta accreta Spectrum (accrete/increta/percreta)
3. Bleeding diathesis
4. Other Causes of Post-Partum Hemorrhage i.e. Uterine atony, Genital tract tears, Retained Products of Conception etc.
5. Serious medical or surgical diseases.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Mean blood loss | 24 hours post procedure
  Mean blood loss within first 24 hours post procedure, was compared in both the groups for outcome measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Awais Qarni, Principal Investigator — Anesthesiologist
Locations (1):
- CMH, Jhelum, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Will only share primary outcome result.